CLINICAL TRIAL: NCT01586208
Title: Refractory Status Epilepticus: Plasmatic Levels Monitorization Utility
Brief Title: Refractory Status Epilepticus Treatment Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Vall d'Hebron (Other); Germans Trias i Pujol Hospital (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Mercè Falip, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NEU-2009-01
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Grand Mal Status Epilepticus; Non-convulsive Status Epilepticus
Keywords: refractory status epilepticus; valproic acid; phenytoin; benzodiazepines; Valproic acid initial dosage in status treatment
MeSH Terms: conditions — Status Epilepticus | interventions — Valproic Acid; Phenytoin; Benzodiazepines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 40mg/kg intial valproate bolus (Active Comparator): Patient receives a 40mg/kg valproate bolus with a maintenance of 1mg/kg/h, after benzodiazepine + phenytoin administration
  Interventions: Drug: valproic acid (VPA)
- 20mg/Kg intial bolus valproate (Active Comparator): Patient receives a 20mg/kg valproate bolus with a maintenance of 1mg/kg/h, after benzodiazepine + phenytoin administration
  Interventions: Drug: valproic acid (VPA)

INTERVENTIONS:
Drug: valproic acid (VPA) — Best dosage at the initial bolus of VPA in patient with satatus epilepticus refractarius (after benzodiazepine + phenytoin treatment)
  Other Names: Valrpoic acid; Phenytoin; Benzodiazepines; Status Epilepticus Refractarius

SUMMARY:
Identify the most effective dose of valproic acid when used in combination with phenytoin for treatment of patients with refractory status epilepticus, which allow a better clinical course and prognosis of the disease.

DETAILED DESCRIPTION:
Phase III Clinical trial, to identify the most effective dose of valproic acid (20mg/kg bolus, 1mg/kg/h maintenance vs 40mg/kg bolus, 2mg/kg/h maintenance) in combination with phenytoin, in patients with refractory status epilepticus.

Multicenter clinical trial, single-blind, prospective, randomized 1:1 assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age who meet the diagnosis of EER seizure, and previously they have been treated according to the clinical protocol at our center status (Diazepam 10mg Clonazepam 1mg and Phenytoin or iv at a dose of 20mg/kg in case persistence of the clinic):

   -Present seizures for at least 30 minutes without regaining awareness among them.
2. Patients ≥ 18 years of age who meet the diagnosis of nonconvulsive EER, and previously they have been treated according to the clinical protocol at our center status (Diazepam 10mg Clonazepam 1mg and Phenytoin or iv at a dose of 20mg/kg in case persistence of the clinic):

   * After submitting an EER seizures that yield clinically performed an EEG that shows SE electricity.
   * Evidence of a non-convulsive SE to perform an EEG of a patient admitted for any cause, either by filing seizures, altered mental status, or any other cause, and to persist after the treatment administered previously discussed.
3. Patients in whom it has obtained the written informed consent by the representative and/or patient, as the case

Exclusion Criteria:

1. Patients with severe cerebral anoxia, when the first EEG evidences a pattern of flare-suppression.
2. Patients who registers PLEDs (periodic epileptic lateralaized Discharges) without clinical seizure activity association to register or without electrical crises.
3. Patients < 18 years of age.
4. Patients in whom there is diagnostic doubt (eg non-convulsive status among and encephalopathy).
5. Pregnant or breastfeeding.
6. Patients with allergy to phenytoin, hydantoin or hypersensitivity to sodium valproate
7. Patients with porphyria
8. Patients with severe liver disease or dysfunction.
9. Patients with heart block or second and third grade sinus bradycardia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
status epilepticus resolution | after 48h treatment administration
  After 48h treatment administration the status epilepticus has to be solved without any other antiepileptic medications

SECONDARY OUTCOMES:
Estimation of pharmacokinetic parameters of valproate (VPA) and phenytoin (PHT) | During 48h post valproate administration
  Estimation of pharmacokinetic parameters of VPA (Cl: clearance, Vd: volume of distribution) and PHT (Vmax: maximum speed of metabolism and Km: plasma concentration at which the rate of metabolism is half the maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Falip, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain